CLINICAL TRIAL: NCT04176991
Title: A Phase 1 Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CTI-1601 Versus Placebo in Subjects With Friedreich's Ataxia
Brief Title: Single Ascending Dose Study of CTI-1601 Versus Placebo in Subjects With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Larimar Therapeutics, Inc. (Industry)
Collaborators: Veristat, Inc. (Other); Metrum Research Group, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-1601-101
Record Dates: First submitted 2019-11-14; First posted 2019-11-26 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTI-1601 (Experimental)
  Interventions: Biological: CTI-1601
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CTI-1601 — CTI-1601 is a recombinant fusion protein and is intended to deliver human frataxin, the protein deficient in Friedreich's ataxia
  Arms: CTI-1601
Biological: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of single ascending doses of CTI-1601 in participants with Friedreich's ataxia

DETAILED DESCRIPTION:
Single Ascending Dose (SAD), Double-Blind, Placebo Controlled Study.

To evaluate the safety and tolerability of single ascending doses of CTI-1601 in subjects with Friedreich's ataxia.

Secondary Objectives:

1. To evaluate the pharmacokinetics (PK) of CTI-1601 following increasing single doses of subcutaneously (SC) administered CTI-1601.
2. To evaluate the pharmacodynamics (PD) of CTI-1601 following increasing single doses of SC administered CTI-1601.

CTI-1601 or Placebo - Dose/Mode of Administration: Single Dose/Subcutaneous

ELIGIBILITY:
Inclusion Criteria:

1. Subject has genetically confirmed Friedreich's ataxia diagnosis, homozygous GAA repeat expansions, with repeat sizing (if available) included on diagnostic report.
2. Subject is male or female, 18 years of age or older at screening.
3. Subject must have a mFARS_neuro score ≥ 20 and be able to traverse a distance of 25 feet with or without some assistive device (cane, walker, crutches, self-propelled wheelchair) and (a) be able to sit upright with thighs together and arms crossed without requiring support on more than two sides; (b) be able to transfer from bed to chair independently or with minimal assistance if, in the opinion of the investigator, the degree of physical disability does not result in undue risk to the subject while participating in the study; and (c) perform basic daily care, such as feeding themselves and personal hygiene, with minimal assistance.
4. Subjects must weigh > 40 kilograms (kg).

Exclusion Criteria:

1. Subjects who are confirmed as compound heterozygous (GAA repeat expansion on only one allele) for Friedreich's ataxia.
2. Subject requires use of amiodarone.
3. Subject used erythropoietin, etravirine, or gamma interferon within 3 months prior to screening.
4. Subject use of investigational drug (other than CTI-1601) or device within 90 days prior to screening.
5. Subject use of daily biotin supplementation that exceeds 30 mcg/day, either as part of a multivitamin or as a standalone supplement, within 7 days prior to study drug administration and/or throughout the entire study.
6. Subject has clinically significant arrhythmia on electrocardiogram (ECG), or evidence of predisposition to significant ventricular arrhythmia on ECG, or evidence of active and unstable coronary artery disease.
7. Male subject who has an ECG QTcF > 450 milliseconds or female subject who has an ECG QTcF > 470 milliseconds.
8. Subject has a screening echocardiogram ejection fraction <45 percent.
9. Subject has a history of aspiration, aspiration pneumonia, or recurrent episodes of pneumonia (greater than or equal to 2 episodes of pneumonia) within the last 12 months.
10. Subjects with known or suspected chronic use of cannabinoid products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | Through study completion, an average of 70 days
  Overall summary of the Participants with Treatment Emergent Adverse Events
Number of Treatment Emergent Adverse Events by System Organ Classification and Preferred Term | Through study completion, an average of 70 days
  Overall summary of Participants with Treatment Emergent Adverse Events by System Organ Classification (MedDRA version 22.0)

SECONDARY OUTCOMES:
Pharmacokinetics - Area under the concentration-time curve after a single dose | Up to 48 hours
  Summary assessment of changes in the area under the concentration-time curve after a single dose
Pharmacokinetics - Maximum observed plasma concentration after a single dose | Up to 48 hours
  Summary assessment of changes in the maximum observed plasma concentration after a single dose
Pharmacokinetics - Time to reach maximum plasma concentration after a single dose | Up to 48 hours
  Summary assessment of changes in time to reach maximum plasma concentration after a single dose
Pharmacokinetics - Area under the concentration-time curve from time 0 to infinity | 48 hours
  Summary assessment of changes in the area under the concentration-time curve from time 0 to infinity
Pharmacokinetics - Area under the concentration-time curve from time 0 to the last measurable time point | 48 hours
  Summary assessment of changes in the Area under the concentration-time curve from time 0 to the last measurable time point
Pharmacokinetics - Apparent total plasma clearance | 48 hours
  Summary assessment of changes in the apparent total plasma clearance
Pharmacokinetics - Terminal half-life estimation | 48 hours
  Summary assessment of changes in the terminal half-life estimation
Pharmacokinetics - Apparent volume of distribution | 48 hours
  Summary assessment of changes in the apparent volume of distribution
Changes from Baseline in Frataxin Levels in Buccal Cells | At baseline and up to 10 days
  Summary assessment of changes in frataxin levels in buccal cells
Changes from Baseline in Frataxin Levels in Whole Blood | At baseline and up to 10 days
  Summary assessment of changes in frataxin levels in whole blood
Changes in Gene Expression Profiling | At baseline and up to 10 days
  Summary assessment of changes in gene expression levels

CONTACTS AND LOCATIONS:
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States

REFERENCES:
- [Background] Koeppen AH. Friedreich's ataxia: pathology, pathogenesis, and molecular genetics. J Neurol Sci. 2011 Apr 15;303(1-2):1-12. doi: 10.1016/j.jns.2011.01.010. PMID 21315377
- [Background] Delatycki MB, Corben LA. Clinical features of Friedreich ataxia. J Child Neurol. 2012 Sep;27(9):1133-7. doi: 10.1177/0883073812448230. Epub 2012 Jun 29. PMID 22752493
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541
- [Background] Plasterer HL, Deutsch EC, Belmonte M, Egan E, Lynch DR, Rusche JR. Development of frataxin gene expression measures for the evaluation of experimental treatments in Friedreich's ataxia. PLoS One. 2013 May 17;8(5):e63958. doi: 10.1371/journal.pone.0063958. Print 2013. PMID 23691127
- See also: Friedreich's Ataxia Research Alliance — http://www.curefa.org/